CLINICAL TRIAL: NCT01264250
Title: A Phase I, Single-centre, Single-blind, Randomised, Placebo-controlled, Single-dose Study to Assess the Safety, Tolerability and Pharmacokinetics After Single Ascending Intravenous Doses of AZD2927 in Healthy Male Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics After Single Ascending Intravenous Doses of AZD2927 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4120C00001
Record Dates: First submitted 2010-12-07; First posted 2010-12-21 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Safety; Tolerability; pharmacokinetics; drug metabolism
MeSH Terms: interventions — AZD2927

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD2927
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2927 — Single dose of AZD2927
  Arms: 1
Drug: Placebo — Single dose of placebo
  Arms: 2

SUMMARY:
In this early phase study, healthy male volunteers will be randomly assigned to one dose of either AZD2927 or placebo. The objective will be to assess the Safety,Tolerability and Pharmacokinetics of AZD2927.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male subjects aged 18 to 45 years inclusive with suitable veins for cannulation or repeated venepuncture
* Male subjects should be willing to use barrier contraception ie, condoms, from the day of dosing until 3 months after dosing with the Investigational Product (IP)
* Have a body mass index (BMI) between 19.0 and 30.0 kg/m2 and weight of at least 50.0 kg and no more than 100.0 kg

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, mental, cardiac, hepatic or renal disorder, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Abnormal vital signs, after 10 minutes supine rest
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of IP
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD2927, at screening | Monitoring of Adverse events, Electrocardiograms, vital signs, safety lab and ophtalmologic variables at screening
Safety and tolerability of AZD2927, day 1 | Monitoring of Adverse events, Electrocardiograms, vital signs, safety lab and ophtalmologic variables on day 1.
Safety and tolerability of AZD2927, day 2 | Monitoring of Adverse events, Electrocardiograms, vital signs and safety lab on day 2.
Safety and tolerability of AZD2927, day 3 | Monitoring of Adverse events, Electrocardiograms, vital signs, and safety lab on day 3.
Safety and tolerability of AZD2927, at follow up | Monitoring of Adverse events, Electrocardiograms, vital signs and safety lab at follow up.

SECONDARY OUTCOMES:
Pharmakokinetic for AZD2927 measured by Cmax, tmax, AUC, t1/2, CL and Vss, day 1 | Pharmacokinetic sampling will be performed day 1
Pharmakokinetic for AZD2927 measured by Cmax, tmax, AUC, t1/2, CL and Vss, day 2 | Pharmacokinetic sampling will be performed day 2
Pharmakokinetic for AZD2927 measured by Cmax, tmax, AUC, t1/2, CL and Vss, day 3 | Pharmacokinetic sampling will be performed day 3

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kühn, MD, Principal Investigator — Quintiles AB; Helen Lunde, MD, Study Director — AstraZeneca; Mirjana Kujacic, MD, Principal Investigator — AstraZeneca
Locations (1):
- Research Site, Uppsala, Sweden